CLINICAL TRIAL: NCT06478043
Title: Phase II Study of AK112 Combined With Irinotecan Liposome in Patients With ES-SCLC Who Progressed on Immune Checkpoint Inhibitors and Chemotherapy.
Brief Title: A Study to Investigate the Efficacy and Safety of Ivonescimab Combined With Irinotecan Liposome as Second-line Regimen for ES-SCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Fan Yun, MD, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-543 (IIT)
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ivonescimab and irinotecan liposome (Experimental): Subjects receive ivonescimab plus irinotecan liposome until progression.
  Interventions: Drug: ivonescimab; Drug: irinotecan liposome

INTERVENTIONS:
Drug: ivonescimab — 20mg/kg, IV, D1, Q3W
  Other Names: AK112
Drug: irinotecan liposome — 56.5mg/m^2, IV, D1, Q2W
  Other Names: Irinotecan liposome injection

SUMMARY:
This is an open-label, single-arm, prospective phase 2 study, evaluating the efficacy and safety of ivonescimab combined with irinotecan liposome for relapsed extensive stage small cell lung cancer, who progressed on PD-(L)1 -based first-line therapy.

DETAILED DESCRIPTION:
Patients will receive ivonescimab at 20mg/kg intravenously, on days 1 of every 21-day cycle and irinotecan liposome 56.5mg/m^2 intravenously, on days 1 of every 14-day cycle. Treatment will be discontnued in case of until the toxicity became intolerable, the investigator determined that there was no further clinical benefit (based on a combination of RECIST V1.1 imaging assessment and clinical status), 24 months of treatment was completed, or the study was withdrawn for other reasons.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old (at the time of inform consent obtained).
2. Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
3. Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Life expectancy of at least 3 months.
6. ES-SCLC who failed first-line platinum-based chemotherapy with checkpoint inhibitors.
7. At least one measurable tumor lesion according to RECIST v1.1.
8. Adequate organ function.
9. All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

1. Patients with other cancer in 5 years.
2. Undergone anti-angiogenic therapy prior to the first dose of study treatment.
3. Evidence and history of severe bleeding tendency.
4. History of severe active autoimmune disease that has required systemic treatment in the past 2 years, severe drug allergy or have known allergy to any component of the study drugs.
5. Active central nervous system (CNS) metastases.
6. Active infection requiring systemic therapy.
7. Current presence of uncontrolled pleural, pericardial, and peritoneal effusions.
8. Active hepatitis B/C, or HIV infection.
9. History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment.
10. History of allogeneic hematopoietic stem cell transplantation or allogeneic organ transplantation.
11. History of alcohol abuse, psychotropic substance abuse or drug abuse.
12. Pregnant or lactating women.
13. Other conditions considered unsuitable for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | Interval between the date of enrollment and the date of death from any cause, up to approximately 2 years
  Objective response rate (ORR) is defined as the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.

SECONDARY OUTCOMES:
Incidence of Grade 3 or higher adverse events (AEs) | Interval between the date of enrollment and the date of death from any cause, up to a maximum of 2 years
  Frequency and severity of adverse events measured according to NCI Common Toxicity Criteria Adverse Event (CTCAE), version 5.0.
Disease control rate (DCR) | Interval between the date of enrollment and the date of death due to any cause , up to a maximum of approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks), based on RECIST v1.1.
Duration of Response (DOR) | Interval between the date of enrollment and the date of death from any cause, up to a maximum of 2 years
  DOR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Progression free survival (PFS) | Interval between the date of enrollment and the date of progressive disease, or death due to any cause (whichever occurs first), up to a maximum of 2 years
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1) assessed by the investigator or death due to any cause (whichever occurs first).
Overall survival (OS) | Interval between the date of enrollment and the date of death from any cause, up to a maximum of 2 years
  OS is the time from the date of randomization or first dosing date to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No